CLINICAL TRIAL: NCT02394639
Title: EEG@HOME (Phase 4 of the Project)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project funding ended before reaching Phase 4.
Sponsor: University Hospital, Ghent (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Pilipili NV (Industry); Imec (Industry)
Responsible Party: Principal Investigator, Neurologie, Prof. dr. Kristl Vonck, University Hospital, Ghent
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: EC/2015/0140
Record Dates: First submitted 2015-02-10; First posted 2015-03-20 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional video-EEG monitoring (Active Comparator): conventional video-EEG monitoring with cup-electrodes and collodion
  Interventions: Other: video-EEG monitoring
- video-EEG monitoring with prototype (Experimental): video-EEG monitoring of 5 hours with EEG-cap with dry electrodes
  Interventions: Other: video-EEG monitoring

INTERVENTIONS:
Other: video-EEG monitoring

SUMMARY:
The goal of this project is the development of an EEG-cap (min. 21 electrodes) with user-friendly active dry electrodes that meets the expectations of the users regarding comfort and esthetics, without losing sight of the functional and technical demands for recording high quality EEG signals. The purpose is to use the EEG-cap to investigate clinical neurological disorders (e.g. epilepsy). The EEG-cap could also be used at home so that hospital admission in the EMU can be avoided for some patients and an increasing number of patients can be examined.

In this stage of the project video-EEG recording with the prototype will be compared to the conventional way (cup-electrodes and collodion) of recording in the EMU.

Minimum 1 - maximum 10 patients with prominent IEDs will be included. After the conventional recording is completed, the patient will undergo a recording of maximum 5 hours with the prototype.

There will be an visual and clinical evaluation of the EEG-signals (blinded) and a technical evaluation of the EEG-signals. User experience and experience of the EEG-technologists will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Epilepsy with on EEG prominent IEDs

Exclusion Criteria:

* /

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
EEG signal quality (visual and clinical) (scale) | 5 hours
EEG signal quality (technical) (signal to noise ratio) | 5 hours
User experience (questionnaire) | 5 hours

SECONDARY OUTCOMES:
EEG-technologist experience (questionnaire) | 5 hours

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - University Hospital, Ghent, Ghent
  - University Hospital, Leuven, Leuven